CLINICAL TRIAL: NCT05376709
Title: A Mixed Methods Study of Nutrition Practice in Cancer Care: Test a Newly-developed Intervention and Establish Frameworks Reflecting Multi-aspects of Eating Behavior Based on Non-Hodgkin Lymphoma Population
Brief Title: A Mixed Methods Study of Nutrition Practice in Cancer Care on Non-Hodgkin Lymphoma Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201810112RIND
Record Dates: First submitted 2020-12-24; First posted 2022-05-17 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-05

CONDITIONS: Lymphoma, B-Cell
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short-Term Calorie Reduction(SCR) (Experimental): To determine the short-term impact of calorie modification on patient outcomes by measuring and comparing the following parameters between two groups a week after starting each R-CHOP cycle: symptoms, hematologic parameters (i.e., erythrocyte-, thrombocytes-, and leucocyte counts), metabolic parameters (i.e., insulin, glucose, insulin growth factor 1), inflammatory response (C-reactive Protein, CRP), and nutrition status (i.e., weight, albumin level, and lean body mass (LBM)).
  Interventions: Dietary Supplement: Short-Term Calorie Reduction
- Control (No Intervention): Participated patients will be recruited and randomized to two groups: comparison group who receive standard care and experimental group who receive the SCR intervention. The standard care at NTUH includes encouraging patients to eat healthy and clean diet (e.g., avoid raw or undercooked food). There are no calorie restriction to the comparison group. The next paragraph describes the SCR intervention for experimental group.

INTERVENTIONS:
Dietary Supplement: Short-Term Calorie Reduction — Align with the R-CHOP regimen, patients in the experimental group will first perform water fast 24 hours before (day 0) and during the first day of R-CHOP (day 1) when they receive Rituximab, Vincristine, Doxorubicin, cyclophosphamide, and prednisolone. On day 2, they will resume normal calorie intake until the day before the next cycle of chemotherapy. While each cycle of R-CHOP takes 21 days, most patients will receive a total of 6-8 cycles over four to six months.
  Arms: Short-Term Calorie Reduction(SCR)

SUMMARY:
The effects of calorie or sugar control on health and disease has been a hot topic. While established evidence has proven the health benefits of long-term calorie restriction, recent preclinical studies show encouraging results of the beneficial effects of short-term fasting on cancer treatment. In particular, short-term calorie control seems to be safe and has the potential to increase cancer cell's sensitivity to chemotherapy whereas protect normal cells from chemotherapy-induced toxicity. More human trials are needed before translating this intervention into clinical practice.

The overall goal of this study is to examine if nutrition status and an intervention of sugar and calorie modification will affect patient outcomes in patients with diffuse large B-Cell lymphoma (DLBCL) receiving chemo therapy which includes Rituximab, Cyclophosphamide, Hydroxydaunomycin, Oncovin, and Prednisone(R-CHOP).

This 5-year research project with three phases will be conducted at National Taiwan University Hospital. The first phase is a case control, observational study. By reviewing electronic charts of patients who (1) were newly diagnosed with DLBCL within the past 5 years, (2) received R-CHOP, (3) were 20-year-old or older at diagnosis, we seek to examine specific aim 1 and 2. About 500 cases are needed in this phase to achieve 80% power. The second phase is a pilot study requiring 50 participants to assess feasibility of the protocol. The third phase is a prospective cohort study in which the safety, feasibility, and effects of a calorie modification protocol are examined (aim 3, 4, and 5), participants will be randomized to experimental and comparison group. While comparison group will receive standard care, experimental group will follow the protocol of calorie modification.

DETAILED DESCRIPTION:
Background. The effects of calorie or sugar control on health and disease has been a hot topic. While established evidence has proven the health benefits of long-term calorie restriction, recent preclinical studies show encouraging results of the beneficial effects of short-term fasting on cancer treatment. In particular, short-term calorie control seems to be safe and has the potential to increase cancer cell's sensitivity to chemotherapy whereas protect normal cells from chemotherapy-induced toxicity. More human trials are needed before translating this intervention into clinical practice.

Study purpose and aims. The overall goal of this study is to examine if nutrition status and an intervention of sugar and calorie modification will affect patient outcomes in patients with diffuse large B-Cell lymphoma (DLBCL) receiving R-CHOP. The specific aims are: (1) to investigate the demographic information and nutrition status (e.g., body mass index, albumin level, fasting sugar, and hyperglycemic episode) of patients with DLBCL before and during R-CHOP; (2) to examine the relationships between nutrition status and treatment outcomes of patients with DLBCL; (3) to evaluate the safety and feasibility of applying the protocol of calorie modification to patients with DLBCL undergoing R-CHOP; (4) to determine the short-term impacts of calorie modification on patient outcomes by measuring and comparing the following parameters between two groups a week after starting each R-CHOP cycle: symptoms, hematologic parameters (i.e., erythrocyte-, thrombocytes-, and leucocyte counts), metabolic parameters (i.e., insulin, glucose, insulin growth factor 1), inflammatory response (C-reactive Protein), and nutrition status (i.e., weight, albumin level, and lean body mass); (5) to determine how calorie modification affects the therapeutic effects of R-CHOP by (a) using positron emission tomography and computed tomography (PET/CT scan) at three time points: before treatment, upon completion of the third cycle, and upon completion of the whole R-CHOP regimen and (b) following up with the progression-free-survival a year post treatment.

Methods and sampling. This 5-year research project with three phases will be conducted at National Taiwan University Hospital. The first phase is a case control, observational study. By reviewing electronic charts of patients who (1) were newly diagnosed with DLBCL within the past 5 years, (2) received R-CHOP, (3) were 20-year-old or older at diagnosis, we seek to examine specific aim 1 and 2. About 500 cases are needed in this phase to achieve 80% power. The second phase is a pilot study requiring 50 participants to assess feasibility of the protocol. The third phase is a prospective cohort study in which the safety, feasibility, and effects of a calorie modification protocol are examined (aim 3, 4, and 5), participants will be randomized to experimental and comparison group. While comparison group will receive standard care, experimental group will follow the protocol of calorie modification. The results of this phase will help finalize the calorie modification protocol and determine the sample size for the third phase which is a larger randomized controlled trial. For phase two and three, the inclusion criteria are patients who are (1) diagnosed with advanced DLBCL, (2) receiving R-CHOP regimen and do not have hypersensitivity reaction, and (3) 20-year-old or older.

Data analysis. Descriptive statistics, Pearson partial correlation, and multiple linear regression will be used to analyze relationship among interested variables. Independent-t test, paired t-test, and Mann-Whitney U test are selected to determine the differences between groups.

Expecting results. The current study is one among the first few translational research programs implementing calorie modification strategies in real practice. It is particularly valuable and innovative in terms of its comprehensive design, extensive scope, and focus of unexplored population. Results of the current study have a great potential to change current nutrition recommendations for cancer patients receiving chemotherapy and enhance evidence-based care.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed with DLBCL
2. Planning to receive R-CHOP regimen
3. 20-year-old or older
4. The targeted sample size is 50 for each group

Exclusion Criteria:

1. Have BMI less than or equal to 18.5
2. Have albumin level lower than 3.4 g/liter
3. History of eating disorders
4. Have difficulties to follow the instructions of calorie modifications due to physiological or psychological condition
5. Have been diagnosed with diabetes mellitus or have physiological or psychological condition that calorie modification may cause negative effect on their physical or psychological status
6. Have special dietary restrictions

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Symptoms at 4 weeks | Baseline and 4 weeks
  European Organization for Research and Treatment of Cancer-Quality of Life Questionnaire core 30. (EORCT-QLQ C30, Taiwan Chinese version) is a reliable and valid tool that a group of experts developed. EORCT-QLQ C30 consists of 30 items and measures patients' functions and symptoms by 4-point Likert scales. Higher scores for symptom scales represent more intense symptoms. Researchers use this measurement to assess the change in symptoms severity before and after chemotherapy.
Change from baseline Quality-of-Life at 4 weeks | Baseline and 4 weeks
  European Organization for Research and Treatment of Cancer-Quality of Life Questionnaire core 30. (EORCT-QLQ C30, Taiwan Chinese version) measures quality-of-life (QoL) by 7-point Likert scales. The minimum and maximum values are 1 and 7, respectively. Higher scores for QoL mean better.
Change from baseline Cell Toxicity at 4 weeks | Baseline and 4 weeks
  To determine the change of short-term impact of calorie modification on patient outcomes by measuring and comparing the hematologic parameters between two groups. The blood sample would be erythrocyte- counts.
Change from baseline Cell Toxicity at 4 weeks | Baseline and 4 weeks
  To determine the change of short-term impact of calorie modification on patient outcomes by measuring and comparing the hematologic parameters between two groups. The blood sample would be thrombocytes- counts.
Change from baseline Cell Toxicity at 4 weeks | Baseline and 4 weeks
  To determine the change of short-term impact of calorie modification on patient outcomes by measuring and comparing the hematologic parameters between two groups. The blood sample would be leucocyte counts.
Change from baseline Cell Metabolism at 4 weeks | Baseline and 4 weeks
  To determine the change of short-term impact of calorie modification on patient outcomes by measuring and comparing the metabolic parameters between two groups. The blood sample would be insulin.
Change from baseline Cell Metabolism at 4 weeks | Baseline and 4 weeks
  To determine the change of short-term impact of calorie modification on patient outcomes by measuring and comparing the metabolic parameters between two groups. The blood sample would be glucose (before meals).
Change from baseline Cell Metabolism at 4 weeks | Baseline and 4 weeks
  To determine the change of short-term impact of calorie modification on patient outcomes by measuring and comparing the metabolic parameters between two groups. The blood sample would be insulin growth factor-1(IGF-1).
Change from baseline Cell Metabolism at 4 weeks | Baseline and 4 weeks
  To determine the change of short-term impact of calorie modification on patient outcomes by measuring and comparing the metabolic parameters between two groups. The blood sample would be prealbumin.
Change from baseline Cell Inflammatory at 4 weeks | Baseline and 4 weeks
  To determine the change of short-term impact of calorie modification on patient outcomes by measuring and comparing the inflammatory parameters between two groups. The blood sample would be like inflammatory response (C-reactive Protein, CRP).
Change from baseline Nutrition Status at 4 weeks | Baseline and 4 weeks
  To determine the short-term impact of calorie modification on patient outcomes by measuring nutrition status with the Inbody S10 Body Water Analyzer machine (i.e., extracellular water).
Change from baseline Nutrition Status at 4 weeks | Baseline and 4 weeks
  To determine the short-term impact of calorie modification on patient outcomes by measuring nutrition status with the Inbody S10 Body Water Analyzer machine (i.e., phase angle)
Change from baseline Nutrition Status at 4 weeks | Baseline and 4 weeks
  To determine the short-term impact of calorie modification on patient outcomes by measuring nutrition status with the Inbody S10 Body Water Analyzer machine (i.e., skeletal muscle mass index, SMI).
Change from baseline PET/CT scan at 18 weeks | Baseline and 18 weeks
  After 6 times chemotherapy, the PET/CT scan will be used to assess the tumor completely response, partially response or progressed compared to the first diagnosed one.

CONTACTS AND LOCATIONS:
Overall Officials: Tai-Chung Huang, MD, Principal Investigator — NTUH
Locations (1):
- NTUH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cathcart P, Craddock C, Stebbing J. Fasting: starving cancer. Lancet Oncol. 2017 Apr;18(4):431. doi: 10.1016/S1470-2045(17)30196-1. No abstract available. PMID 28368246